CLINICAL TRIAL: NCT06226701
Title: EFFECT OF CRYOLIPOLSIS IN HORMONAL PROFILE AND MENSTRUAL REGULARITY IN OBESE WOMEN WITH PCOS
Brief Title: EFFECT OF CRYOLIPOLYSIS ON HORMONAL PROFILE AND MENSTRUAL REGULARITYIN OBESE WITH PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sabrin Mohamed Taha Abdelwahab (Other)
Responsible Party: Sponsor-Investigator, Sabrin Mohamed Taha Abdelwahab, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.tRec/012/004763
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Obese Women With PCOS
Keywords: obesity, pcos ,cryolipolysis
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Impact of cryolipolsis on hormonal Profile in obese women with Pcps
Who Masked: Participant, Care Provider
Masking Description: Double (participant,outcomes assessed random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impact of cryolipolsis on hormonal profile in obese women with pcos (Experimental): The patients will receive cryolipolysis session in abdomen for 45minute ,session every two week and 1200kcal diet and exercise for 3 months
  Interventions: Device: Cryolipolysis device
- Impact of cryolipolysis in hormonal profile in obese women with pcos (Experimental): All patient will receive same diet 1200kcal diet ,and exercise for 3 months
  Interventions: Device: Cryolipolysis device

INTERVENTIONS:
Device: Cryolipolysis device — -Cryolipolysis device
  1max cool shaping device ( inform china korean technology).Is used for fat lipolysis ,with no harm to the skin.The device consist of Cool sculptor applicator head , cool gel pad its alarge gel pad it should be adherent to the area to be treated before applying the cool sculptor applicator to protect the skin from bruising or ecchymosis. The device uses vacuum suction which can be adjusted according to the patient tolerance. Duration of session 45min at each of treatment session ,1session every 2weeks for 3months.
  Other Names: max freeze device

SUMMARY:
The effecting study to determine the impact of cryolipolysis on obese women with pcos

DETAILED DESCRIPTION:
Polycystic ovary syndrome(PCOS) is the most common endocrine disorder in women of reproductive age. Women with this syndrome may have infrequent menstrual periods or amenorrhea and excess androgen levels. The ovaries develop numerous small follicles and fail to ovulate on a regular basis, with subsequent subfertility in those women that wish to conceive.The etiology of PCOS is unclear. Early diagnosis and treatment may reduce the risk of long-term complications such as type 2 diabetes and heart disease ,PCOS affects 5-20% of women of reproductive age worldwide. The condition is characterized by hyperandrogenism, ovulatory dysfunction and polycystic ovarian morphology (PCOM) with excessive androgen production by the ovaries being a key feature of PCOS. PCOS is classified into four separate phenotypes (A-D), according to the presence or absence of three characteristics: hyperandrogenism (either biochemical or clinical), ovulatory dysfunction and polycystic ovarian morphology. Only phenotype A requires all three features of PCOS to be present. The various diagnostic criteria currently available for PCOS include a greater or fewer number of PCOS phenotypes. AE-PCOS, Androgen Excess-PCOS Society; NIH, National Institutes of Health ,the trial made on 2group ,control group and study group for 3 months

ELIGIBILITY:
Inclusion Criteria:

All patient age from 18to 30 Waist hip ratio >.9

Exclusion Criteria:

* thyroid disorders. Hepatic diseases. Skin or bleeding disorders. Chronic disease or illnessCardiovascular and pulmonary disease,Cancer diseases., Renal failure disease. Recent surgery. hose with pacemakers or surgical implants. Musculoskeletal problems that would limit WBV.Raynaud's phenomenon. A rare condition in which cold temperatures can impede blood flow to the fingers and toes. Other conditions that pose a risk include,Pregnancy or breast-feeding,Inflammatory skin disorders,Skin conditions caused by immune system disorders, such as eczema or psoriasis

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Weight | Up to 3months
  the scale will asses the weight of patient
Hormones | 3months
  blood sample will take by lab before and after treatment

SECONDARY OUTCOMES:
waist hip ratio | 3months
  waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement (W⁄H). For example, a person with a 75 cm waist and 95 cm hips (or a 30-inch waist and 38-inch hips) has WHR of about 0.79.

CONTACTS AND LOCATIONS:
Locations (1):
- Sabrin mohamed taha abdelwahab, Bilbeis, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes